CLINICAL TRIAL: NCT06714201
Title: CUrrent Practices of Intensive Care for the Management of Acute Respiratory Distress Syndrome in EurOpe.
Acronym: CUPIDO
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Università degli Studi di Trento (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Genova (Other); University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Markus Haar, Specialist in Internal Medicine, University of Hamburg-Eppendorf
Other Study IDs: UKE-KIM-MH-001
Record Dates: First submitted 2024-11-19; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: ARDS; Prone position; ECMO; ECCO2R; vvECMO; vv-ECMO; Mechanical Ventilation; Tidal volume
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study seeks to gain a comprehensive understanding of current ARDS management practices across European ICUs, with a particular focus on the use of LTV and PP therapy, which have been shown to improve outcomes in ARDS patients. The primary objectives focus on evaluating how LTV and PP are implemented across different institutions, while secondary objectives encompass a broader assessment of other ARDS treatment strategies. These include mechanical ventilation approaches, including PEEP titration, the use of NMBAs, and advanced extra-corporal therapies like ECMO and extracorporeal carbon dioxide removal (ECCO2R). Additionally, the study will explore diagnostic methods and decision-making processes that guide ARDS management in diverse clinical settings.

DETAILED DESCRIPTION:
This is a cross-sectional survey designed to collect data on the current practices of ARDS management in ICUs across Europe. The survey will be administered electronically, allowing for the efficient collection of responses from a broad and diverse group of healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

• Healthcare professionals (physicians and nurses) who are currently employed in an ICU that treats ARDS patients and are actively involved in their management.

Exclusion Criteria:

• There are no specific exclusion criteria for this study, as the aim is to gather as broad a range of perspectives and practices as possible from ICUs treating ARDS patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of healthcare professionals directly involved in the management of ARDS patients in European ICUs. This includes a multidisciplinary group of:
  * Physicians at various levels of responsibility and expertise, such as medical directors, senior physicians, attending consultants, and assistant physicians.
  * ICU nurses actively participating in the care and management of ARDS patients. To ensure broad and representative participation, we will collaborate with national representatives who are engaged in ARDS research. These representatives will be instrumental in leveraging their professional networks to facilitate access to local clinicians working in ICUs. By doing so, we aim to capture a diverse and comprehensive range of clinical practices and insights into the management of ARDS across Europe.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of ICUs utilising prone positioning for ARDS patients. | Survey period (December 2024 - March 2025)
  This measure evaluates the adoption of prone positioning therapy across ICUs in Europe, capturing variations in its implementation for ARDS patients.
PaO2/FiO2 threshold for starting prone positioning. | Survey period (December 2024 - March 2025)
  This measure represants a categorical variable and captures the clinical thresholds for initiating prone positioning, based on the PaO2/FiO2 ratio.
Distribution of the extent of prone positioning used in participating ICUs. | Survey period (December 2024 - March 2025).
  This measure categorises the extent of prone positioning in ARDS patients based on typical positioning angles (e.g., 135°, 180°) and reports the proportion of ICUs using each category.
  Unit of Measure: Percentage of ICUs per category (e.g., 135°, 180°).
Mean duration per prone positioning cycles. | Survey period (December 2024 - March 2025)
  Evaluates the typical duration of individual prone positioning cycle. Unit of Measure: Hours per cycle
Mean minimum number of prone position cycles. | Survey period (December 2024 - March 2025)
  Evaluates the minumum number of prone position cycles per patient, regardless of therapy response.
  Unit of Measure: number of cycles (count)
Commonly reported criteria for ending prone positioning therapy. | Survey period (December 2024 - March 2025)
  Assesses clinical and physiological criteria used to determine the cessation of prone positioning, such as oxygenation improvements or complications. Descriptive frequencies of criteria.
Proportion of ICUs adhering to tidal volume restrictions | Survey period (December 2024 - March 2025)
  Measures the compliance of ICUs with evidence-based lung-protective ventilation strategies in ARDS patients, focusing on tidal volume settings.
  Unit of Measure: Percentage.
Mean tidal volumes used for mild, moderate, and severe ARDS. | Survey period (December 2024 - March 2025)
  Captures variations in tidal volume settings based on the severity of ARDS, aiming to identify trends in lung-protective strategies.
  Unit of Measure: mL/kg predicted body weight.

SECONDARY OUTCOMES:
Proportion of ICUs using volume-controlled vs pressure-controlled ventilation. | Survey period (December 2024 - March 2025)
  Examines ICU preferences for mechanical ventilation modes, highlighting trends in volume-controlled and pressure-controlled ventilation strategies.
  Unit of Measure: Percentage.
Types of PEEP titration methods and recruitment manoeuvres. | Survey period (December 2024 - March 2025)
  Evaluates PEEP titration strategies, including the use of recruitment manoeuvres and their clinical application in ARDS management.
  Unit of Measure: Percentage.
Proportion of ICUs using NMBAs for ARDS patients. | Survey period (December 2024 - March 2025).
  Captures the frequency of NMBA use and its role in facilitating lung-protective ventilation in ARDS management.
  Unit of Measure: Percentage.
Frequency of corticosteroid and nitric oxide use. | Survey period (December 2024 - March 2025)
  Investigates the use of adjunct pharmacological therapies in ARDS management, focusing on corticosteroids and inhaled nitric oxide.
  Unit of Measure: Percentage.
Proportion of ICUs with ECMO/ECCO2R availability and implementation. | Survey period (December 2024 - March 2025).
  Assesses the availability of advanced extracorporeal therapies and their integration into ARDS treatment protocols.
  Unit of Measure: Percentage.
Variation in prone position extent by country. | Survey period (December 2024 - March 2025).
  Explores the influence of country of medical practice on the extent of prone position being performed (full prone position vs. parital prone position).
  Unit of Measure: Proportions

IPD SHARING:
Plan to Share IPD: No